CLINICAL TRIAL: NCT07252076
Title: PRetreatment MRI for OCcult Liver Metastasis Assessment In Pancreatic Ductal adenocarcinoMa. An International Multicentric, Prospective, Diagnostic Accuracy Trial
Brief Title: PRetreatment MRI for OCcult Liver Metastasis Assessment In Pancreatic Ductal adenocarcinoMa
Acronym: PROCLAIM
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.ChirGen.25.03
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample will be taken from patients included in the study and stored prior to surgery for possible future investigations into biological markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Contrast-enhanced MRI and DWI sequences — Assessment of the accuracy of contrast-enhanced MRI and DWI sequences in detecting liver metastases in PDAC that are not identified on CT and evaluation of the clinical impact of adding this imaging modality to the diagnostic algorithm in this specific patient population.

SUMMARY:
Pancreatic cancer has a low survival rate largely due to late diagnosis and undetected liver metastases. Computed tomography (CT), the standard diagnostic tool, often misses occult metastases that are later discovered during surgery. Recent studies suggest that magnetic resonance imaging (MRI), especially with diffusion-weighted imaging (DWI), can better detect very small liver metastases and help avoid unnecessary surgery. However, MRI is not yet widely used in routine practice due to limited evidence and its selective application. This study proposes incorporating contrast-enhanced MRI and DWI into the diagnostic workflow to improve diagnostic accuracy and guide more effective treatment decisions for patients with pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is a deadly disease with a low five-year survival rate, mainly due to late diagnosis and distant metastases, particularly to the liver. Computed tomography (CT) is the conventional diagnostic method, but it does not always detect hidden liver metastases, which are often only identified during surgery. Recent studies suggest that the use of magnetic resonance imaging (MRI), especially with diffusion-weighted imaging (DWI) sequences, could improve the detection of occult liver metastases, even those smaller than one centimeter, and thus influence treatment decisions, reducing unnecessary surgery.

However, the adoption of MRI as standard practice is not yet widespread, due to the lack of evidence and its limited use in specific situations. This study proposes integrating contrast-enhanced MRI and DWI into the diagnostic protocol to refine diagnostic accuracy and therapeutic choices, with the aim of optimizing treatment and survival in patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years of age.
* Patients with a new cytological or histological diagnosis of PDAC.
* A CT scan demonstrating pancreatic disease and meeting the minimum criteria for the imaging assessment of pancreatic gland tumors (see section 4.6, study procedures).
* An MRI performed no later than 3 weeks after the CT scan, also meeting the minimum radiological criteria (see section 4.6, study procedures).
* No prior treatment for pancreatic disease.
* Patients able to receive and understand the study information and to provide written informed consent duly signed by both the patient and the investigator.

Exclusion Criteria:

* Signs of metastatic disease on the initial CT scan (hepatic, pulmonary, distant lymph node, peritoneal carcinomatosis, or other organ involvement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received a histopathological diagnosis of pancreatic ductal adenocarcinoma and have undergone contrast-enhanced CT without evidence of metastatic disease, defined as the presence of suspicious lesions in the liver, lungs, distant lymph nodes, peritoneum, or other organs.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients | Through study completion, an average of 18 months
  Percentage of patients in whom MEOs will be detected on MRI in the intention-to-image population after negative CT for secondary lesions.

SECONDARY OUTCOMES:
Identification of the target sequences | Through study completion, an average of 18 months
  Identification of the most accurate sequences for detecting MEOs on MRI

OTHER OUTCOMES:
Predictive model creation | Through study completion, an average of 18 months
  Based on the results of the first objective, a predictive model will be created, to identify patients at high risk of MEO.

CONTACTS AND LOCATIONS:
Locations (1):
- SC Chirurgia Generale, Alessandria, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No